CLINICAL TRIAL: NCT07216105
Title: A Phase 1, Open-Label Study of FT836, an Off-the-Shelf CAR T-Cell Therapy, With or Without Chemotherapy and/or Monoclonal Antibodies, in Participants With Advanced Solid Tumors
Brief Title: FT836 With or Without Chemotherapy and/or Monoclonal Antibodies, in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT836-101
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer; Breast Cancer; Ovarian Cancer; Endometrial Carcinoma; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC, NSCLC, CRC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel; Cetuximab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Regimen A ( FT836) (Experimental): Participants receive FT836 monotherapy
  Interventions: Drug: FT836
- Regimen B ( Paclitaxel + FT836) (Experimental): Participants receive Paclitaxel chemotherapy followed by FT836
  Interventions: Drug: FT836; Drug: Paclitaxel
- Regimen C ( Cetuximab + FT836) (Experimental): Participants receive FT836 combined with cetuximab
  Interventions: Drug: FT836; Drug: Cetuximab
- Regimen D ( Paclitaxel + Cetuximab + FT836) (Experimental): Participants receive Paclitaxel chemotherapy followed by FT836 combined with cetuximab
  Interventions: Drug: FT836; Drug: Paclitaxel; Drug: Cetuximab
- Regimen E ( Trastuzumab + FT836)) (Experimental): Participants receive FT836 combined with trastuzumab
  Interventions: Drug: FT836; Drug: Trastuzumab
- Regimen F ( Paclitaxel + Trastuzumab + FT836) (Experimental): Participants receive Paclitaxel chemotherapy followed by FT836 combined with trastuzumab
  Interventions: Drug: FT836; Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: FT836 — FT836 drug product is administered as an intravenous infusion on multiple days schedule at treatment cycle.
  Other Names: 836
Drug: Paclitaxel — IV infusion ; 80 mg/m2 QW; Days -21, -14, and -7
  Other Names: Taxol
  Arms: Regimen B ( Paclitaxel + FT836); Regimen D ( Paclitaxel + Cetuximab + FT836); Regimen F ( Paclitaxel + Trastuzumab + FT836)
Drug: Cetuximab — Cetuximab administration will begin on Day -4 at the recommended initial dose of 400 mg/m2 as a 120-minute IV infusion
  Other Names: Erbitux
  Arms: Regimen C ( Cetuximab + FT836); Regimen D ( Paclitaxel + Cetuximab + FT836)
Drug: Trastuzumab — trastuzumab administration will begin on Day -4 at an initial dose of 4 mg/kg as a 90-minute IV infusion.
  Other Names: Herceptin
  Arms: Regimen E ( Trastuzumab + FT836)); Regimen F ( Paclitaxel + Trastuzumab + FT836)

SUMMARY:
This is a phase 1 study of FT836 administered in participants with advanced solid tumors. The primary objectives of the study are to evaluate the safety and tolerability of FT836 with or without paclitaxel and/or trastuzumab or cetuximab, and to determine the recommended phase 2 dose (RP2D) of FT836 in combination with trastuzumab or cetuximab; each objective will be assessed with or without paclitaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* For all regimens, disease that is not amenable to curative therapy and that has relapsed or progressed following at least one line of prior systemic therapy.
* Evidence of adequate organ function as determined by all of the following:

  * Absolute neutrophil count (ANC) >1000/µL without growth factor support within 7 days prior to start of first study intervention
  * Platelet count ≥75,000/µL without transfusion support within 14 days prior to start of first study intervention
  * Estimated creatinine clearance ≥50 mL/minute by Cockcroft-Gault method or other standard institutional method
  * Total bilirubin ≤1.5 × upper limit of normal (ULN); for participants with documented Gilbert syndrome, total bilirubin must be ≤3 ×ULN
  * Aspartate transaminase (AST) ≤3 × ULN or alanine transaminase (ALT) ≤3 × ULN; in participants with documented liver metastases, AST or ALT ≤5 × ULN
  * Alkaline phosphatase (ALP) ≤2.5 × ULN; in participants with documented liver or bone metastases, ALP ≤5 × ULN
  * Oxygen saturation >90% on room air
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Presence of measurable disease by RECIST, v1.1 assessed within 28 days prior to start of first study intervention.
* Presence of baseline safely accessible lesions of adequate size for on-treatment biopsies (exceptions for lesion size may be granted with medical monitor approval) and participant willingness to undergo protocol prescribed on-treatment biopsies.

Exclusion Criteria:

* Clinically significant cardiovascular disease including any of the following: uncontrolled/ unstable cardiac arrhythmias, myocardial infarction within 6 months prior to start of first study intervention, unstable angina or congestive heart failure of New York Heart Association (NYHA) Grade 2 or higher, or cardiac ejection fraction <50%.
* Receipt of any biological therapy, chemotherapy, investigational therapy, or radiation therapy within 2 weeks or five half-lives prior to start of fifirst study intervention, whichever is shorter.
* Known active central nervous system (CNS) involvement by malignancy. Participants with prior CNS involvement from their malignancy must have completed effective treatment of their CNS disease with no symptoms of disease in the absence of steroid treatment and at least stable findings on relevant CNS imaging and no evidence of leptomeningeal disease for at least 4 weeks prior to study enrollment.
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions within 6 months prior to study enrollment.
* Currently receiving or likely to require systemic immunosuppressive therapy (e.g., prednisone ≥5 mg daily) for any reason from start of first study intervention to Day 29 with the exception of corticosteroids as a premedication for chemotherapy side effects per institutional standard of care or as mandated by the protocol.
* Any history of Grade ≥3 immune-related AE or Grade ≥2 eye toxicity attributed to prior cancer immunotherapy, other than endocrinopathy managed with replacement therapy or asymptomatic elevation of serum amylase or lipase.
* Grade ≥2 peripheral neuropathy limiting instrumental activities of daily living.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | From Day 1 through Day 29 of Cycle 1( each cycle is 56 days)
  The number of participants experiencing ≥1 DLT will be reported.
Severity of DLTs | From Day 1 through Day 29 of Cycle 1( each cycle is 56 days)
  The severity of DLTs will be determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, v5.0).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months
  Participants will be classified into the following tumor response categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or not evaluable (NE) per RECIST v1.1. The best overall response (BOR) will be summarized for the efficacy evaluable population. ORR is defined as the percentage of participants who achieve a PR or better during the study prior to any subsequent off-protocol anti-cancer therapy.
Duration of Response (DOR) | Up to approximately 24 months
  The DOR is defined as the time from first objective response to disease progression or death from any cause.
Progression-Free Survival (PFS) | Up to approximately 24 months
  PFS is defined as the time from first study intervention to progressive disease or death from any cause.
Overall Survival (OS) | Up to approximately 24 months
  OS is defined as the time from first dose of study intervention to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Dempster, Study Director — Fate Therapeutics
Locations (3):
- United States (3):
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - M. D. Anderson Cancer Center, Houston, Texas